CLINICAL TRIAL: NCT00830869
Title: An Open-Label, Dose Escalation, Phase 1 Study of IXAZOMIB (MLN9708), a Second-Generation Proteasome Inhibitor, in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: A Phase 1 Study of IXAZOMIB in Adult Patients With Advanced Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16001; U1111-1206-2180 (Other: WHO)
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Advanced Non-hematologic Malignancies
Keywords: Drug therapy
MeSH Terms: interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1: Ixazomib 0.125 milligram per square meter (mg/m^2) (Experimental): Ixazomib (MLN9708) 0.125 mg/m^2, injection, intravenously (IV), once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
  Interventions: Drug: IXAZOMIB
- Part 1: Ixazomib 0.25 mg/m^2 (Experimental): Ixazomib (MLN9708) 0.25 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
  Interventions: Drug: IXAZOMIB
- Part 1: Ixazomib 0.5 mg/m^2 (Experimental): Ixazomib (MLN9708) 0.5 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
  Interventions: Drug: IXAZOMIB
- Part 1: Ixazomib 1 mg/m^2 (Experimental): Ixazomib (MLN9708) 1 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
  Interventions: Drug: IXAZOMIB
- Part 1: Ixazomib 1.33 mg/m^2 (Experimental): Ixazomib (MLN9708) 1.33 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
  Interventions: Drug: IXAZOMIB
- Part 1: Ixazomib 1.76 mg/m^2 (Experimental): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
  Interventions: Drug: IXAZOMIB
- Part 1: Ixazomib 2.34 mg/m^2 (Experimental): Ixazomib (MLN9708) 2.34 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study. Once the MTD will be established, participants with NSCLC, Head and Neck Cancer (H&N), Soft Tissue Sarcoma (STC) or Prostate Cancer (PC) will be included in MTD disease expanded cohort. An additional tumor pharmacodynamics expansion cohort (TPEC) will enroll participants with any type of solid tumor that can be biopsied for tissue analysis before and after treatment with ixazomib.
  Interventions: Drug: IXAZOMIB
- Part 2:Ixazomib 1.76 mg/m^2-NSCLC (Experimental): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with NSCLC during Part 2 of the study.
  Interventions: Drug: IXAZOMIB
- Part 2: Ixazomib 1.76 mg/m^2-H&N (Experimental): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with H&N during Part 2 of the study.
  Interventions: Drug: IXAZOMIB
- Part 2: Ixazomib 1.76 mg/m^2-STC (Experimental): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with STC during Part 2 of the study.
  Interventions: Drug: IXAZOMIB
- Part 2: Ixazomib 1.76 mg/m^2-PC (Experimental): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with PC during Part 2 of the study.
  Interventions: Drug: IXAZOMIB
- Part 2: Ixazomib 1.76 mg/m^2-TPEC (Experimental): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with various types of solid tumors suitable for biopsy in tumor pharmacodynamic expansion cohort (TPEC) during Part 2 of the study.
  Interventions: Drug: IXAZOMIB

INTERVENTIONS:
Drug: IXAZOMIB — All participants will receive IXAZOMIB IV injection on Days 1, 4, 8, and 11 of each treatment cycle followed by a rest period of 10 days.
  The first stage of the study will be initiated at a starting dose of 0.125 mg/m^2. Subsequent doses will increase until a maximum tolerated dose (MTD) is established.

SUMMARY:
This is an open-label, multicenter, phase 1, dose escalation study of IXAZOMIB. The primary purpose of this study is to determine the safety profile, establish the maximum tolerated dose, and inform the phase 2 dose of IXAZOMIB administered intravenously in participants with nonhematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

1. Male or female participants 18 years or older.
2. Eastern Cooperative Oncology Group performance status 0-2.
3. A diagnosis of a nonhematologic malignancy for which standard treatment is no longer effective. In the expanded cohort, enrollment will be limited to participants with a diagnosis of NSCLC, H&N cancer (squamous cell cancer), STS, or PC.
4. Suitable venous access for pharmacokinetic (PK) and pharmacodynamic evaluations.
5. Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.

   Male participants who agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.
6. Voluntary written consent must be obtained.
7. Adequate clinical laboratory values during the screening period.
8. In the escalation portion of the study, radiographically or clinically evaluable tumor was required, but measurable disease as defined by response evaluation criteria in solid tumors (RECIST) criteria was not required. In the MTD disease expansion cohorts and the TPEC, clinically measurable disease as defined by RECIST criteria was required for evaluation of NSCLC, H&N cancer, and STS. Prostate specific antigen (PSA) alone was acceptable for evaluation of PC.
9. For participants in the TPEC, tumor tissue that, in the opinion of the investigator, could have been safely biopsied using a core needle.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Peripheral neuropathy greater than or equal to (>=) Grade 2.
2. Female participants who are lactating or have a positive serum pregnancy test during the screening period.
3. Major surgery within 14 days before the first dose of treatment.
4. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before the first dose of study treatment.
5. Life-threatening illness unrelated to cancer.
6. Diarrhea greater than (>) Grade 1 based on the National Cancer Institute Common Terminology .Criteria for Adverse Events (NCI CTCAE) categorization.
7. Systemic antineoplastic therapy / or radiotherapy within 21 days before the first dose of study treatment.
8. Systemic treatment with prohibited medications.
9. Participant has symptomatic brain metastasis.
10. Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or myocardial infarction within the past 6 months.
11. QTc >470 milliseconds (msec) on a 12-lead electrocardiogram (ECG) obtained during the screening period.
12. Known human immunodeficiency virus (HIV), hepatitis B or hepatitis C positive.
13. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
14. Treatment with any investigational products within 28 days before the first dose of study treatment.
15. For participants in the TPEC and participants in the MTD disease expansion cohorts who gave informed consent to undergo tumor biopsy, ongoing anticoagulant therapy (example, aspirin, clopidogrel [Plavix ®], warfarin, or heparin) that cannot be held to permit tumor biopsy .
16. Known allergy to boron or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-03-02 (Actual); Primary Completion 2012-04-20 (Actual); Study Completion 2012-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- United States (6):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Washington- Seattle Cancer Care, Seattle, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States and Canada from 02 March 2009 to 20 April 2012.
Pre-assignment Details: Participants with diagnosis of nonhematologic malignancies were enrolled in 1 of the 2 parts, Part 1: Dose escalation to determine maximum tolerated dose (MTD), and Part 2: Expansion at MTD in 5 expansion cohorts.
Groups:
- Part 1: Ixazomib 0.125 mg/m^2: Ixazomib (MLN9708) 0.125 milligram per square meter (mg/m^2), injection, intravenously (IV), once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
- Part 1: Ixazomib 2.34 mg/m^2: Ixazomib (MLN9708) 2.34 mg/m^2, injection, IV, once on Day 1, 4, 8 and 11 followed by 10 days of rest in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity during Part 1 of the study.
- Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with NSCLC during Part 2 of the study.
- Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with H&N during Part 2 of the study.
- Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with STC during Part 2 of the study.
- Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC): Ixazomib (MLN9708) 1.76 mg/m^2, injection, IV, once on Day 1, 4, 8, and 11 followed by 10 days of rest period in 21-day treatment cycles for a maximum of 12 cycles, or until progressive disease or unacceptable toxicity in participants with PC during Part 2 of the study.
Period: Period 1: Part 1
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Started | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Symptomatic deterioration | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 1 | 6 | 4 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Part 2
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 22 | 20 | 11 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 22 | 20 | 11 | 20
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 2 | 2 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 1 | 4
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 11 | 12 | 8 | 15
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of ixazomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC | Total
Number analyzed (Participants) | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 20 | 22 | 20 | 11 | 20 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 55.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 69.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 55.1 (10.71) | 59.8 (14.22) | 62.3 (10.98) | 64.7 (10.79) | 58.6 (11.50) | 55.1 (9.99) | 55.0 (9.43) | 63.1 (5.49) | 57.6 (11.24) | 57.8 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 5 | 3 | 3 | 0 | 10 | 4 | 12 | 0 | 10 | 50
  Male | 0 | 0 | 0 | 2 | 1 | 3 | 3 | 10 | 18 | 8 | 11 | 10 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 0 | 1 | 1 | 6 | 1 | 6 | 3 | 17 | 19 | 16 | 9 | 18 | 97
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 3 | 3 | 3 | 1 | 2 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 7 | 14
  White | 1 | 1 | 1 | 7 | 4 | 5 | 2 | 17 | 18 | 17 | 10 | 12 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 0 | 6 | 4 | 5 | 3 | 16 | 20 | 19 | 11 | 20 | 106
  Canada | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 2 | 1 | 0 | 0 | 10
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 163.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 173.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 156.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 168.9 (8.19) | 163.3 (9.54) | 167.8 (11.44) | 178.3 (5.69) | 170.0 (7.61) | 173.8 (9.11) | 164.2 (11.54) | 178.3 (6.72) | 171.4 (9.23) | 170.4 (9.91)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 79.70 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 65.50 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 64.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 73.37 (20.517) | 66.33 (16.589) | 70.90 (21.377) | 85.47 (14.086) | 70.87 (11.160) | 69.00 (12.448) | 74.06 (19.650) | 94.20 (14.321) | 91.44 (30.468) | 77.17 (20.794)
Body surface area [Mean (Standard Deviation); unit: square meter (m^2)] | 1.90 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1.80 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1.70 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1.83 (0.298) | 1.73 (0.250) | 1.82 (0.331) | 2.03 (0.153) | 1.82 (0.151) | 1.82 (0.197) | 1.84 (0.276) | 2.15 (0.181) | 2.08 (0.383) | 1.90 (0.282)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicity (DLT)
Description: Toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0. DLT is any of following related to ixazomib:Grade (GR) 4 neutropenia (absolute neutrophil count<500 cells/cubic meter[cells/mm^3])for>7 days; GR 3 neutropenia with coincident fever and/or infection; GR 4 thrombocytopenia (platelets <25,000 cells/mm3)for>7 days; GR 3 thrombocytopenia with clinically significant bleeding; Platelet count<10,000 cells/mm3; GR 3 peripheral neuropathy;>=GR 3 nausea/emesis in absence of optimal antiemetic therapy; >=GR 3 diarrhoea in absence of optimal supportive therapy;GR 3 QTc prolongation noted on average of 3 electrocardiograms (ECGs);>=GR 3 nonhematological toxicity except GR 3 arthralgia/myalgia or GR 3 fatigue for<1 week; Delay in initiation of subsequent therapy cycle by>7 days due to treatment-related toxicity Other>=GR 2 nonhematological toxicity that opinion of investigator, requires discontinuation of therapy with Ixazomib.
Time Frame: Part 1: Cycle 1 Day 1 up to Cycle 1 Day 21
Population: The DLT population included all participants who received all Cycle 1 doses of ixazomib and who had completed Cycle 1. If Cycle 1 was interrupted by a DLT, the participant was included in this population.
Measure: Number; unit: participants
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 7 | 4 | 6 | 3
participants | 0 | 0 | 0 | 1 | 0 | 1 | 3

2. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Event (SAEs)
Time Frame: Part 1: Cycle 1 Day 1 up to Cycle 10 Day 41; Part 2: Cycle 1 Day 1 up to Cycle 12 Day 41
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 20 | 22 | 20 | 11 | 20
participants
  TEAEs | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 20 | 22 | 19 | 11 | 20
  SAEs | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 9 | 10 | 7 | 6 | 11

3. Primary Outcome: Number of Participants With Clinically Significant TEAEs Related to Laboratory Abnormalities
Time Frame: Day 1 up to 30 days after last dose of study drug (Cycle 12 Day 41)
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 20 | 22 | 20 | 11 | 20
participants
  Liver function analyses | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
  Renal function analyses | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 1
  Tissue enzyme analyses notelsewhereclassified(NEC) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Red blood cell analyses | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Platelet analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
  Mineral and electrolyte analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Metabolism tests NEC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Urinalysis NEC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Thrombocytopenias | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 8 | 12 | 8 | 6 | 14
  Anaemias NEC | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 3 | 3 | 6 | 1 | 4
  Leukopenias NEC | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 7
  Neutropenias | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2
  Leukocytoses NEC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Marrow depression and hypoplastic anaemias | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Thrombocytoses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sodium imbalance | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 6 | 3
  Hyperglycaemic conditions NEC | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
  Potassium imbalance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
  Calcium metabolism disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
  Magnesium metabolism disorders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Disorders of purine metabolism | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Metabolic acidoses (excluding diabetic acidoses) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Phosphorus metabolism disorders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Protein metabolism disorders NEC | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation and bleeding analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital sign measurements included diastolic and systolic blood pressure, heart rate, weight and oral temperature.
Time Frame: Day 1 up to 30 days after last dose of study drug (Cycle 12 Day 41)
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 1 | 1 | 1 | 7 | 4 | 6 | 3 | 20 | 22 | 20 | 11 | 20
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Part 1: AUC (0-72): Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours Post-dose for Ixazomib
Description: AUC (0-72) is a measure of the area under the plasma concentration-time curve from time 0 to 72 hours post-dose for ixazomib.
Time Frame: Part 1: Cycle 1 Days 1 and 11: pre-dose and at multiple time points (up to 72 hours) post-dose
Population: PK analysis population where data at specified time points was available,defined as participants in dose escalation phase who received protocol-specified dosing in Cycle 1 without dose reductions/interruptions, did not receive excluded concomitant medications in Cycle 1,had sufficient concentration-time data to permit estimation of PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 4 | 6 | 1
nanogram*hour per milliliter (ng*hr/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 4 | 4 | 6 | 1
  Cycle 1 Day 1 |  |  | 91.6 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 191.87 (40.211) | 391.46 (92.446) | 522.74 (120.122) | 620.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.
  Cycle 1 Day 11: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 5 | 1
  Cycle 1 Day 11 |  | 60.9 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 301.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 579.91 (246.505) | 1161.92 (424.774) | 1542.64 (454.015) | 3800.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

6. Secondary Outcome: Part 1: C0: Initial Plasma Concentration After Bolus Intravenous Administration
Description: C0 is the plasma drug concentration at time zero following bolus intravenous injection.
Time Frame: Part 1: Cycle 1 Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose; Cycle 1 Day 11 pre-dose and at multiple time points (up to 264 hours) post-dose
Population: PK analysis population where data at specified time points was available, defined as participants in dose escalation phase who received protocol-specified dosing in Cycle 1 without dose reductions/interruptions,did not receive excluded concomitant medications in Cycle 1,had sufficient concentration-time data to permit estimation of PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per mililiter (ng/mL)
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 4 | 6 | 1
nanogram per mililiter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 6 | 1
  Cycle 1 Day 1 | 15.1 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 82.5 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 192.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 346.70 (170.208) | 366.16 (146.167) | 579.54 (210.672) | 901.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.
  Cycle 1 Day 11: number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 5 | 1
  Cycle 1 Day 11 | 27.1 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 69.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 83.8 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 272.57 (64.044) | 390.08 (209.538) | 648.97 (597.508) | 869.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

7. Secondary Outcome: Part 1: Rac: Accumulation Ratio for Ixazomib
Description: Rac was estimated as the ratio of AUC (0-72) on Day 11 and AUC (0-72) on Day 1. AUC (0-72) is the area under the plasma concentration-time curve from time 0 to 72 hours post-dose.
Time Frame: Cycle 1 Day 11 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: PK analysis population defined as participants in dose escalation phase who received protocol-specified dosing in Cycle 1 without dose reductions/interruptions,did not receive excluded concomitant medications in Cycle 1,had sufficient concentration-time data to permit estimation of PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 5 | 1
ratio | 2.210 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 5.160 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 3.290 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 2.996 (1.5948) | 2.831 (0.7228) | 3.086 (0.4998) | 6.130 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

8. Secondary Outcome: Part 1: Terminal Phase Elimination Half-life (T1/2) for Ixazomib
Description: T1/2 is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Part 1: Cycle 1 Day 11 pre-dose and at multiple time points (up to 264 hours) post-dose
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 5 | 1
hours |  |  |  | 171.90 (38.070) | 144.69 (27.647) | 104.84 (39.646) | 90.80 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

9. Secondary Outcome: Part 1: E Max: Maximum Observed Effect for Ixazomib
Description: E max is the maximum inhibition of 20S proteasome activity in whole blood.
Time Frame: as for outcome 6
Population: PD analysis population where baseline/post-baseline assessments was available, defined as participants in dose escalation phase who received protocol-specified dosing in Cycle 1 without dose reductions/interruptions,did not receive any excluded concomitant medications in Cycle 1,had sufficient effect-time data to permit estimation of PD parameters.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 4 | 6 | 1
percentage of inhibition
  Cycle 1 Day 1 | 7.70 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 17.90 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 28.20 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 35.22 (8.592) | 46.73 (9.424) | 62.20 (9.862) | 67.40 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.
  Cycle 1 Day 11: number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 5 | 1
  Cycle 1 Day 11 | 4.50 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 10.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 46.10 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 39.33 (8.868) | 54.30 (4.058) | 61.90 (9.042) | 70.40 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

10. Secondary Outcome: Part 1: TEmax: Time to Maximum Observed Effect (Emax) for Ixazomib
Description: TEmax is the time to reach the Emax, equal to time (hours) to Emax.
Time Frame: Part 1: Cycle 1 Days 1 and 11 pre-dose and at multiple time points (up to 72 hours) post-dose; Cycle 1 Day 11 pre-dose and at multiple time points (up to 264 hours) post-dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 4 | 6 | 1
hour
  Cycle 1 Day 1 | 1.000 [1.00 to 1.00] | 0.100 [0.10 to 0.10] | 0.250 [0.25 to 0.25] | 0.100 [0.08 to 0.10] | 0.250 [0.10 to 0.25] | 0.080 [0.07 to 0.10] | 0.080 [0.08 to 0.08]
  Cycle 1 Day 11: number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 5 | 1
  Cycle 1 Day 11 | 24.000 [24.00 to 24.00] | 0.080 [0.08 to 0.08] | 0.100 [0.10 to 0.10] | 0.110 [0.10 to 0.12] | 0.080 [0.08 to 0.10] | 0.120 [0.08 to 0.18] | 0.100 [0.10 to 0.10]

11. Secondary Outcome: Number of Participants With Best Overall Response
Description: Best overall response for a participant is best observed post-baseline disease response as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 criteria. Complete Response (CR): disappearance of all target lesions, non-target lesions and normalization of tumor marker level. Partial Response (PR): at least 30% decrease in sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the baseline smallest sum of longest diameter; persistence of 1 or more non-target lesion(s) or maintenance of tumor marker level above normal limits. Progressive disease: at least 20% increase in the sum of the longest diameter of target lesions, taking as reference the baseline smallest sum of longest diameter or appearance of 1 or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Day 18 up to Day 21 of each cycle (Part 1: up to Cycle 10; Part 2: up to Cycle 12)
Population: The response-evaluable population included all participants who received at least 1 cycle of ixazomib treatment, had measurable disease at baseline, and had at least 1 postbaseline response assessment.
Measure: Number; unit: participants
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 1 | 1 | 1 | 6 | 3 | 5 | 2 | 15 | 14 | 16 | 11 | 17
participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  SD | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 5 | 5 | 8 | 3 | 3
  Progressive disease | 1 | 0 | 1 | 5 | 3 | 3 | 0 | 10 | 8 | 8 | 7 | 14

12. Secondary Outcome: Part 2: Ixazomib Concentration in Postdose Clinical Tumor Samples in Ixazomib 1.76 mg/m^2-TPEC
Description: The average data of Days 1 and 4 of Cycle 1 was reported.
Time Frame: Cycle 1 Days 1 and 4: Predose and (from 4-20 hours) post-dose
Population: The tumor PK analysis set where Day 1 and 4 assessment were available. The tumor PK and PD analysis population includes all participants who provided a baseline tumor biopsy sample and 1 post-baseline tumor biopsy sample on Day 1 or Day 4.
Measure: Mean (Standard Deviation); unit: nanogram per gram (ng/g)
Arm/Group | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 10
nanogram per gram (ng/g) | 525 (342)

13. Secondary Outcome: 20S Proteasome Activity of Ixazomib in the Tumor Tissue
Time Frame: Cycle 1 Days 1 and 4 pre-dose and at multiple time points (up to 2 hours of tumor biopsy) post-dose
Population: This outcome measure was not analyzed due to lack of tumor activity data.
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Expression of Biomarker (ATF-3) in Tumor Tissue
Time Frame: Cycle 1 Days 1 and 4 pre-dose and at multiple time points (up to 2 hours of tumor biopsy) post-dose
Population: This outcome measure was not analyzed due to lack of tumor activity data.
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to Part 1: Cycle 10 Day 41, Part 2: Cycle 12 Day 41)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Ixazomib 0.125 mg/m^2 | Part 1: Ixazomib 0.25 mg/m^2 | Part 1: Ixazomib 0.5 mg/m^2 | Part 1: Ixazomib 1 mg/m^2 | Part 1: Ixazomib 1.33 mg/m^2 | Part 1: Ixazomib 1.76 mg/m^2 | Part 1: Ixazomib 2.34 mg/m^2 | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) | Part 2: Ixazomib 1.76 mg/m^2-TPEC
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 1/7 | 1/4 | 0/6 | 1/3 | 0/20 | 2/22 | 1/20 | 0/11 | 1/20
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 0/1 | 1/7 | 1/4 | 4/6 | 3/3 | 9/20 | 10/22 | 7/20 | 6/11 | 11/20
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 7/7 | 4/4 | 6/6 | 3/3 | 20/20 | 22/22 | 20/20 | 11/11 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ixazomib 0.125 mg/m^2 (N=1) | Part 1: Ixazomib 0.25 mg/m^2 (N=1) | Part 1: Ixazomib 0.5 mg/m^2 (N=1) | Part 1: Ixazomib 1 mg/m^2 (N=7) | Part 1: Ixazomib 1.33 mg/m^2 (N=4) | Part 1: Ixazomib 1.76 mg/m^2 (N=6) | Part 1: Ixazomib 2.34 mg/m^2 (N=3) | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) (N=20) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) (N=22) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) (N=20) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) (N=11) | Part 2: Ixazomib 1.76 mg/m^2-TPEC (N=20)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ixazomib 0.125 mg/m^2 (N=1) | Part 1: Ixazomib 0.25 mg/m^2 (N=1) | Part 1: Ixazomib 0.5 mg/m^2 (N=1) | Part 1: Ixazomib 1 mg/m^2 (N=7) | Part 1: Ixazomib 1.33 mg/m^2 (N=4) | Part 1: Ixazomib 1.76 mg/m^2 (N=6) | Part 1: Ixazomib 2.34 mg/m^2 (N=3) | Part 2:Ixazomib 1.76 mg/m^2-Non-small Cell Lung Cancer(NSCLC) (N=20) | Part 2: Ixazomib 1.76 mg/m^2-Head and Neck Cancer (H&N) (N=22) | Part 2: Ixazomib 1.76 mg/m^2-Soft Tissue Sarcoma (STC) (N=20) | Part 2: Ixazomib 1.76 mg/m^2-Prostate Cancer (PC) (N=11) | Part 2: Ixazomib 1.76 mg/m^2-TPEC (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 3 | 3 | 7 | 8 | 5 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 3 | 2 | 3 | 1 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 5 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 4 | 3 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 2 | 2 | 1 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 1 | 4 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 7 | 3 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 4 | 7 | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Horner's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phantom pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | 2 | 2 | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 3 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 7 | 3 | 5 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 2 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory depth decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 5 | 3 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 3 | 2 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 5 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disorder of orbit (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Auricular perichondritis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Auricular swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.